CLINICAL TRIAL: NCT01675973
Title: A Phase 1, Parallel-group, Open-label, Multiple-dose Study to Assess the Pharmacokinetics, Safety, and Tolerability of Ranolazine ER in Subjects With Severe Renal Impairment as Compared to Healthy Subjects With Normal Renal Function
Brief Title: A Phase 1 Study to Assess the Effect of Severe Renal Impairment on the Pharmacokinetics, as Well as Safety/Tolerability, of Ranolazine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study met stopping criteria specified within protocol.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-259-0112
Record Dates: First submitted 2012-07-26; First posted 2012-08-30 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Severe Renal Impairment
Keywords: Ranolazine; renal impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — Ranolazine

ARMS (2):
- Subjects with severe renal impairment (Experimental): Cohort B (subjects with severe RI): Approximately 10 subjects will be enrolled to obtain approximately 8 evaluable subjects.
  Interventions: Drug: RANEXA
- Subjects with normal renal function (Experimental): Cohort A (healthy subjects with normal renal function): Approximately 10 subjects will be enrolled to obtain approximately 8 evaluable subjects.
  Interventions: Drug: RANEXA

INTERVENTIONS:
Drug: RANEXA — 500mg BID up to 1000mg BID

SUMMARY:
The purpose of this study is to assess the effect of severe renal impairment on the steady-state PK, as well as safety and tolerability, of ranolazine, compared to subjects with normal renal function.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the effects of severe renal impairment (RI) on the steady-state pharmacokinetics (PK) of ranolazine and key metabolites. The secondary objective of this study is to assess the safety and tolerability of multiple oral doses of ranolazine in subjects with severe RI.

ELIGIBILITY:
Inclusion criteria (All Cohorts):

* Males and females, 18 to 75 years old, inclusive
* Body mass index (BMI) 18 to 40 kg/m2, inclusive, at Screening
* Females of child-bearing potential must have a negative pregnancy test at Screening and on Day -1 (Cohort A) or Day -6 (Cohort B) and must agree to use highly effective contraception methods from Screening throughout the duration of the Treatment Period and for 14 days following the last dose of study drug

Inclusion criteria (Cohort A [Healthy subjects with normal renal function] only):

* Estimated creatinine clearance (CLCR), according to the Cockcroft-Gault (C-G) equation, ≥ 90 mL/min at Screening
* Age, BMI, and sex comparable to those of subjects of Cohort B
* Good health status as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations

Inclusion criteria (Cohort B, Severe RI):

* Diagnosis of CKD
* Estimated glomerular filtration rate (eGFR), according to the Modification of Diet in Renal Disease (MDRD) equation, < 30 mL/min/1.73 m2 (and not receiving dialysis)
* Stable medication dose and dosing regimen for treatment of the complications of renal disease or other concomitant chronic illnesses for at least 2 weeks prior to study drug administration

Exclusion Criteria:

Exclusion criteria (All Cohorts):

* History of uncontrolled or unstable cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease
* Current or recent (within 3 months) gastrointestinal (GI) disease or any GI surgery that could impact absorption of study drug
* Any major surgery within 4 weeks of dosing with study drug
* Donation of blood or plasma to a blood bank or in a clinical study (except a screening visit) within 4 weeks of dosing with study drug
* Blood transfusion within 4 weeks of dosing with study drug
* Consumption of > 14 alcoholic drinks per week, or more than 4 alcoholic drinks on any one day
* History of regular use of tobacco- or nicotine-containing products in excess of 10 cigarettes per day or equivalent
* History of substance abuse within 12 months prior to Screening
* Positive drug screen
* Positive alcohol test
* Clinically significant history of hepatic disease
* QTcF interval > 480 msec at Screening or Day -6 (for Cohort B) or Day -1 (for Cohort A)
* History of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia, or torsade de pointes
* Known hypersensitivity or previous intolerance to ranolazine or any of its excipients
* Treatment with selected medications
* Pregnancy or lactation
* Other condition(s) that, in the opinion of the Investigator, would prevent compliance with the study protocol

Exclusion criteria (Cohort A [Healthy subjects with normal renal function] only):

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations
* Hemoglobin < 12 g/dL for males, < 11 g/dL for females at Screening
* Any prescription and over-the-counter medications, including herbal products

Exclusion criteria (Cohort B, Severe RI):

* Any clinical, ECG, and laboratory findings beyond those which are consistent with the degree of renal dysfunction
* History of or anticipated near-term need for renal transplant (within 3 months)
* History of hemodialysis or peritoneal dialysis within 1 year prior to Screening, or anticipated need for hemodialysis or peritoneal dialysis during the study
* History of acute renal failure or nephrotic syndrome within 1 year prior to Screening
* History of diabetic ketoacidosis
* History of severe hypoglycemia
* Other condition(s) that, in the opinion of the Investigator, would prevent compliance with the study protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration vs time curve over the dosing interval at steady state (AUCtau) and Maximum observed plasma concentration at steady-state (Cmax) | Day 7 for Cohorts A & B, and Day -1 for Cohort B only.
  * Maximum observed plasma ranolazine concentration at steady-state (Cmax) [Time frame: 0, 1, 2, 3, 4, 6, 8, 10, and 12 hours post-dose on Day 7 for Cohort A and Days -1 and 7 for Cohort B]
  * Area under the plasma ranolazine concentration versus time curve over the dosing interval at steady state (AUCtau) [Time frame: 0, 1, 2, 3, 4, 6, 8, 10, and 12 hours post-dose on Day 7 for Cohort A and Days -1 and 7 for Cohort B]

SECONDARY OUTCOMES:
Number of subjects with AEs | From Day -5 for Cohort B or Day 1 for Cohort A through the 14-day follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States